CLINICAL TRIAL: NCT05083429
Title: Replication of the POET-COPD Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-POET-COPD
Record Dates: First submitted 2021-09-20; First posted 2021-10-19 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate; Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Salmeterol inhaler: Reference group
  Interventions: Drug: Salmeterol
- Tiotropium: Exposure group
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Salmeterol — Salmeterol inhaler dispensing claim is used as the reference
  Groups: Salmeterol inhaler
Drug: Tiotropium — Tiotropium dispensing claim is used as the reference
  Groups: Tiotropium

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal than 40: days [0,0]
* Diagnosis of COPD: days [-All Data, 0]
* History of at least 1 COPD exacerbation within the past year requiring treatment with antibiotics and/or systemic steroids and/or requiring hospitalization: days [-365, -28]

Exclusion Criteria:

* Patients with 3 diagnosis of asthma: days [-180, 0]
* Patients with current severe cardiovascular disorders (Heart Transplantation, LVAD/Implantable heart, Pulmonary hypertension/other pulmonary disease) and use of systemic corticosteroid medication at unstable doses: days [-365, 0]
* Patients with any respiratory infection (Acute respiratory infections, pneumonia and influenza) or COPD exacerbation: days [-28, 0]
* Exclude use of salmeterol or tiotropium containing inhaler use [-180, 0]

Ages: 40 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive pulmonary disease (COPD)
Sampling Method: Non-Probability Sample
Enrollment: 8716 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
Time to first COPD exacerbation | [Time Frame: To censoring or study completion, up to 365 days]
  Time to first COPD exacerbation

SECONDARY OUTCOMES:
All-cause death | [Time Frame: To censoring or study completion, up to 365 days]
  All-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT05083429/Prot_SAP_000.pdf